CLINICAL TRIAL: NCT01830959
Title: Use of Roflumilast to Prevent Exacerbations in Fibrotic Sarcoidosis Patients (REFS)
Acronym: REFS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: The Cleveland Clinic (Other); University of Pittsburgh (Other); University of Illinois at Chicago (Other); Henry Ford Health System (Other); Albany Medical College (Other)
Responsible Party: Principal Investigator, Robert P Baughman, Professor of Medicine, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REFS-1; WIRB Pr #: 20130426 (Other: WIRB)
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Sarcoidosis
Keywords: Sarcoidosis, fibrosis, bronchiectasis
MeSH Terms: conditions — Sarcoidosis; Fibrosis; Bronchiectasis | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Roflumilast (Experimental): Roflumilast
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — Roflumilast
  Other Names: Daliresp
  Arms: Roflumilast
Drug: Placebo — Placebo one a day
  Arms: Placebo

SUMMARY:
Pulmonary sarcoidosis patients with fibrosis often develop recurrent episodes of bronchitis. These can lead to worsening of disease for both the short and long term.

Roflumilast has been shown to reduce the number of acute bronchitis episodes in patients with COPD.

Drugs similar to Roflumilast have been shown to help sarcoidosis. The current study is to determine if Roflumilast will reduce number of episodes of bronchitis and help fibrotic sarcoidosis.

DETAILED DESCRIPTION:
This will be a multicenter, double blind, placebo controlled study. Patients would be randomized 1:1 to receive either roflumilast 500 mcg per day or placebo added to their current treatment regimen for twelve months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sarcoidosis as defined by the American Thoracic Society criteria
2. Patients with an FEV1/FVC ratio of less than 80%
3. Patients with fibrosis on chest x-ray and/or high resolution CT scan.
4. Patients have had at least two exacerbations of their sarcoidosis in the prior year. An exacerbation is defined as an acute event requiring increase of prednisone with or without use of antibiotics.
5. Patients must be on a stable dose of corticosteroids and other agents for their sarcoidosis at least 4 weeks prior to first visit.
6. For patients on prednisone alone, the dose has to be the equivalent of 5 mg prednisone a day. For those on other immunosuppressants, they can be on any dose of prednisone.
7. Patients must be between ages of 18 and 70 years of age.
8. Willing to take prednisone at increased dosage for exacerbations of their sarcoidosis.
9. Patients must be able to provide written informed consent to participate in the study.

Exclusion Criteria:

1. Patients with known hypersensitivity to theophylline or pentoxifylline will not be eligible. Patients with dose dependent nausea from these drugs may still participate in the trial.
2. Patients will not be able to take theophylline or pentoxifylline during the time of the study. They will be allowed to take drugs for sarcoidosis including prednisone, methotrexate, azathioprine, leflunomide, hydroxychloroquine, thalidomide, infliximab, adalimumab, and rituximab.
3. Patients with serum creatinine of greater than 3 mg/dL
4. Patients with moderate or severe liver disease as defined Child Pugh class 3 or 4.
5. Patients with unstable cardiac disease
6. Patients with non cutaneous malignancy treated in the past two years.
7. Patients unable to complete the questionnaires and six minute walks detailed in the study.Women of child bearing potential unable to use adequate birth control as determined by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-05 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Reduction in number of episodes of acute exacerbation | one year
  Collect number of episodes of exacerbtion in one year

SECONDARY OUTCOMES:
Change in FVC | one year
  Changes in FVC over time of the study
Changes in quality of life | One year
  Measure QOL using Sarcoidosis health question, fatigue assessment score, SGRQ, SF-36 Leicester cough questionnaire

OTHER OUTCOMES:
Safety | one year
  recard adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Baughman, MD, Study Chair — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Baughman RP, Judson MA, Culver DA, Birring SS, Parambil J, Zeigler J, Lower EE. Roflumilast (Daliresp(R)) to reduce acute pulmonary events in fibrotic sarcoidosis: a multi-center, double blind, placebo controlled, randomized clinical trial. Sarcoidosis Vasc Diffuse Lung Dis. 2021;38(3):e2021035. doi: 10.36141/svdld.v38i3.11684. Epub 2021 Sep 30. PMID 34744427